CLINICAL TRIAL: NCT00238004
Title: The Low HDL On Six Weeks Statin Therapy (LOW) Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Craigavon Area Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-001690-26
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: HDL Cholesterol; Coronary Arteriosclerosis; Lipoproteins
Keywords: Niacin
MeSH Terms: conditions — Coronary Artery Disease | interventions — Niacin

INTERVENTIONS:
Drug: Nicotinic acid

SUMMARY:
Abnormal blood cholesterol levels increase the risk of developing, or dying from heart disease. It is well recognised that if "harmful" LDL cholesterol is high, and "protective" HDL cholesterol is low, this risk is increased. Drugs called statins are routinely used in patients with heart disease, are well tolerated, and decrease the harmful LDL cholesterol levels. However, statins only increase protective HDL cholesterol to a small extent. Some patients may thus benefit from additional medication to increase protective HDL-cholesterol further. One of the most effective drugs which can do this is nicotinic acid. This drug is well established having been available for over 30 years. Previous use has been limited by facial flushing in a large percentage of patients receiving the drug. However a new formulation called Niaspan is now available which is associated with much less flushing. Although many patients will have transient flushing, it is estimated that only 1 patient out of every 20 receiving the drug will have to discontinue treatment. We therefore propose, in patients with coronary artery disease and low HDL cholesterol despite being on a statin, to study the effect of Niaspan on HDL cholesterol and other lipid parameters, and to assess its tolerability.

DETAILED DESCRIPTION:
Objective: To assess, in patients with coronary heart disease and low HDL-cholesterol, the efficacy and tolerability of Niaspan as an adjunct to statin therapy in clinical practice.

Background: Despite the clear reduction in mortality and cardiovascular morbidity associated with reduction of LDL cholesterol (LDL-C) by statin therapy, a sizeable proportion of patients remain at risk of subsequent adverse cardiac events [1-3]. It is clear that in some patients, further risk reduction may be obtained by addressing other elements of the lipid profile. In particular, sub-analysis of the Framingham study has shown that for any given level of LDL-C, the risk of coronary heart disease events decreased with increasing HDL cholesterol (HDL-C) levels [4]. In addition, the adverse cardiac risk associated with elevated triglycerides is predominantly seen in patients with low HDL-C levels [5]. The protective effect of HDL-C appears predominantly mediated via reverse cholesterol transport. In this process, excess cholesterol in cell membranes is transferred to HDL-C in the peripheral tissues, cholesterol is converted to cholesteryl ester in HDL-C by lecithin:cholesterol acyltransferase (LCAT), the newly synthesized cholesteryl ester is transported from HDL-C to lower density lipoproteins by the action of cholesteryl ester transfer protein (CETP) and finally, the cholesterol is removed from plasma by hepatic clearance of plasma lipoproteins. Of the available licensed lipid lowering agents, nicotinic acid has the greatest potential for raising HDL-C, in addition to giving favourable reductions in LDL-C, triglycerides, lipoprotein (a), apolipoprotein B-100 and elevation of Apolipoprotein A-1.

Early studies with nicotinic acid confirmed its efficacy in improving cardiac outcomes. The Coronary Drug Project [6], studied 8341 men with previous MI. A 26% reduction in non fatal MI and 24% reduction in cerebrovascular events was reported after 6 years follow up [6] and an 11% reduction in mortality after 15 years follow up [7]. The Stockholm Ischemic Heart Disease Secondary Prevention Study [8] compared niacin plus clofibrate vs. placebo in 555 post MI survivors and after 5 years reported a 26% reduction in overall mortality (p<0.05) and 36% reduction in CHD mortality (p<0.01). In the current era, statin therapy is considered mandatory for patients with confirmed coronary artery disease [3]. However, nicotinic acid appeared safe and efficacious in combination with statin therapy as demonstrated in the more recent HDL Atherosclerosis Treatment Study (HATS) [9], where the frequency of the composite end point (death, MI, stroke, or revascularization) was reduced from 24% with placebo to 3% with simvastatin-niacin therapy. While flushing was previously a use limiting factor with the immediate release nicotinic acid (niacin), a new extended release preparation (Niaspan) has reduced the incidence of use limiting flushing to <6%. Several studies demonstrate the ability of Niaspan to improve HDL levels, either as monotherapy [10,11], or in addition to statin therapy [12]. To date the safety and efficacy of Niaspan has not been studied in a placebo controlled manner, in a group of patients with coronary artery disease already on statin therapy.

Study population: Patients will be recruited primarily from the cardiology wards of Craigavon Cardiac Centre, Craigavon Area Hospital.

Inclusion criteria:

1. Persisting low HDL-C (<0.9mmol/l) on a full lipid profile result (which for inpatients should have been taken <24 hours after admission).
2. Objective diagnosis of coronary heart disease (previous biomarker proven MI, positive stress test, angiogram with at least one >50% diameter stenosis)
3. Established for at least 6 weeks on a "maintenance" dose of statin therapy (defined as Pravastatin 40mg, Simvastatin 40mg or Atorvastatin ≥10mg). The dose and type of statin should not be altered during the study period
4. Absence of concurrent major systemic illness (particularly liver or renal failure, or hypo or hyperthyroidism)

Exclusion criteria:

1. Previous use of Niaspan or other non-statin lipid lowering agent within the previous 12 weeks
2. Contraindications to Niaspan therapy
3. Participation in another medical trial within the previous 30days
4. Failure to obtain informed consent

Study Design: To be considered as a pilot study. Patients will be prospectively randomized, in a double blind fashion with 1:1 ratio, to receive Niaspan or to an otherwise identical placebo, with doses titrated according to the clinical response. The primary outcome measure will be the number of patients achieving target HDL-C levels (defined as HDL-C >1.0mmol/l in males or >1.29mmol/l in females) after completion of the study protocol while taking Niaspan compared with placebo. The final HDL-C blood sample for comparative analysis between groups will be taken at week 11, or at week 15, if the HDL-C target had not been reached by week 11. Given the HDL-C inclusion criteria of <0.9mmol/l, assuming a least difference to detect of 0.09mmol, and allowing for study drop outs, 30 patients per group will have >90% power to detect this difference as statistically significant. Analysis by intention to treat will be made by an independent samples T test.

References

1. Randomised trial of cholesterol lowering in 4444 patients with coronary heart disease: the Scandinavian Simvastatin Survival Study (4S) Lancet 1994;344:1383-9.
2. LIPID Study Investigators. Long-term risk stratification for survivors of acute coronary syndromes. Results from the Long-term Intervention with Pravastatin in Ischemic Disease (LIPID) Study. J Am Coll Cardiol 2001;38:56-63.
3. MRC/BHF Heart Protection Study of cholesterol-lowering with simvastatin in 5963 people with diabetes: a randomised placebo-controlled trial. Lancet 2003;361:2005-16.
4. Castelli WP, Anderson K, Wilson PW, Levy D. Lipids and risk of coronary heart disease. The Framingham Study. Ann Epidemiol 1992;2(1-2):23-8.
5. Gordon T, Castelli WP, Hjortland MC, Kannel WB, Dawber TR. High density lipoprotein as a protective factor against coronary heart disease. The Framingham Study. Am J Med 1977;62:707-14
6. Gans DJ. Coronary Drug Project JAMA 1975;234:21-2
7. Canner PL, Berge KG, Wenger NK, Stamler J, Friedman L, Prineas RJ, Friedewald W. Fifteen year mortality in Coronary Drug Project patients: long-term benefit with niacin. J Am Coll Cardiol 1986;8:1245-55.
8. Carlson LA, Rosenhamer G. Reduction of mortality in the Stockholm Ischaemic Heart Disease Secondary Prevention Study by combined treatment with clofibrate and nicotinic acid. Acta Med Scand. 1988;223(5):405-18.
9. Brown BG, Zhao XQ, Chait A, Fisher LD, Cheung MC, Morse JS, Dowdy AA, Marino EK, Bolson EL, Alaupovic P, Frohlich J, Albers JJ. Simvastatin and niacin, antioxidant vitamins, or the combination for the prevention of coronary disease. N Engl J Med. 2001 Nov 29;345(22):1583-92.
10. Capuzzi DM, Guyton JR, Morgan JM, Goldberg AC, Kreisberg RA, Brusco OA, Brody J. Efficacy and safety of an extended-release niacin (Niaspan): a long-term study. Am J Cardiol 1998;8274U-81U.
11. Morgan JM, Capuzzi DM, Guyton JR. A new extended-release niacin (Niaspan): efficacy, tolerability, and safety in hypercholesterolemic patients. Am J Cardiol 1998;82:29U-34U.
12. Wolfe ML, Vartanian SF, Ross JL, Bansavich LL, Mohler ER 3rd, Meagher E, Friedrich CA, Rader DJ. Safety and effectiveness of Niaspan when added sequentially to a statin for treatment of dyslipidemia. Am J Cardiol 2001;87(4):476-9, A7.
13. Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation 2002;106(25):3143-421.
14. Mosca L, et al. AHA scientific statement. Evidence-based guidelines for cardiovascular disease prevention in women. Circulation. 2004;109:672-693.

ELIGIBILITY:
Inclusion Criteria:

* Persisting low HDL-C (<0.9mmol/l) on a full lipid profile result (which for inpatients should have been taken <24 hours after admission).
* Objective diagnosis of coronary heart disease (previous biomarker proven MI, positive stress test, angiogram with at least one >50% diameter stenosis)
* Established for at least 6 weeks on a "maintenance" dose of statin therapy (defined as Pravastatin 40mg, Simvastatin 40mg or Atorvastatin ≥10mg). The dose and type of statin should not be altered during the study period
* Absence of concurrent major systemic illness (particularly liver or renal failure, or hypo or hyperthyroidism)

Exclusion Criteria:

* Previous use of Niaspan or other non-statin lipid lowering agent within the previous 12 weeks
* Contraindications to Niaspan therapy
* Participation in another medical trial within the previous 30days
* Failure to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-11

PRIMARY OUTCOMES:
Number of patients achieving target HDL-C levels (defined as HDL-C >1.0mmol/l in males or >1.29mmol/l in females) after completion of the study protocol

SECONDARY OUTCOMES:
Incidence and severity of flushing

CONTACTS AND LOCATIONS:
Overall Officials: I Menown, MD FRCP, Principal Investigator — Craigavon Area Hospital
Locations (1):
- Craigavon Cardiac Centre, Craigavon, United Kingdom